CLINICAL TRIAL: NCT04297215
Title: Pragmatic Randomized Controlled Multi Center Trial Comparing the Effectiveness of Antibacterial Therapeutic Clothing Based on Silver or Chitosan as Compared With Non-antibacterial Therapeutic Clothing in Patients With Moderate to Severe Atopic Dermatitis
Brief Title: The Effectiveness of Antibacterial Therapeutic Clothing Based on Silver or Chitosan as Compared With Non-antibacterial Therapeutic Clothing in Patients With Moderate to Severe Atopic Dermatitis
Acronym: ABC project
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Erasmus Medical Center (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); UMC Utrecht (Other); St. Antonius Hospital (Other); ZonMw: The Netherlands Organisation for Health Research and Development (Other); BAP Medical (Unknown); D&M B.V. (Unknown); DeclaCare (Unknown); University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Suzanne G.M.A. Pasmans, Principal Investigator, MD, PhD Professor, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Erasmus MC 108933
Record Dates: First submitted 2019-09-04; First posted 2020-03-05 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Atopic Dermatitis
Keywords: Atopic dermatitis; Staphylococcus aureus; Therapeutical clothing; Anti-infective agents
MeSH Terms: conditions — Dermatitis, Atopic; Staphylococcal Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Placebo Comparator): This group will receive therapeutic clothing without antimicrobial agents
  Interventions: Device: Binamed® therapeutic clothing without antimicrobial agents
- Chitosan group (Active Comparator): This group will receive antimicrobial therapeutic clothing based on chitosan
  Interventions: Device: DermaCura® Chitosan based antimicrobial therapeutic clothing
- Silver group (Active Comparator): This group will receive antimicrobial clothing based on silver.
  Interventions: Device: Binamed® silver based antimicrobial therapeutic clothing

INTERVENTIONS:
Device: DermaCura® Chitosan based antimicrobial therapeutic clothing — DermaCura® antimicrobial therapeutic clothing (D&M) consists of 98% TENCEL® and 2% elastane. 1% chitosan has been added to TENCEL®
  The therapeutic clothing is to be worn at night during the 12-month intervention period and if needed during the day. Usual care including application of emollients, corticosteroid ointments or creams only if needed and/or antihistamines is continued, with standardized steroid ointments and treatment regimens for comparability purposes.
  Arms: Chitosan group
Device: Binamed® silver based antimicrobial therapeutic clothing — The Binamed® antimicrobial therapeutic clothing (BAP Medical) consists of micro-modal, lycra and woven silver filaments as antibacterial agent.
  The therapeutic clothing is to be worn at night during the 12-month intervention period and if needed during the day. Usual care including application of emollients, corticosteroid ointments or creams only if needed and/or antihistamines is continued, with standardized steroid ointments and treatment regimens for comparability purposes.
  Arms: Silver group
Device: Binamed® therapeutic clothing without antimicrobial agents — The Binamed® therapeutic clothing without antimicriobial agents (BAP Medical) is therapeutic clothing made of micro-modal and lycra. Micro-madal is a semi-synthetic wood cellulose fiber. This fiber has a high strength hand elasticity, a high moisture-permeability and feels soft. Lycra ensures an optimal fit on the skin.
  The therapeutic clothing is to be worn at night during the 12-month intervention period and if needed during the day. Usual care including application of emollients, corticosteroid ointments or creams only if needed and/or antihistamines is continued, with standardized steroid ointments and treatment regimens for comparability purposes.
  Arms: Control group

SUMMARY:
Since 2000 therapeutic clothing or functional textiles based on silver or chitosan as antibacterial agents were introduced as therapeutics of atopic dermatitis (AD). These agents aim to reduce skin colonization with Staphylococcus (S.) aureus. S. aureus induces further dysregulation of the inflammatory process and increased colonization with S. aureus is correlated with increased AD severity. Based on the theoretical mode of action and clinical experience, we assume a higher effectiveness of antimicrobial therapeutic clothing compared to control therapeutic clothing on reducing AD severity. The goal of this study is to assess the effectiveness of antibacterial clothing based on silver or chitosan on the doctor-reported AD severity in patients with moderate to severe AD. Secondary goals are to retrieve information about the effect of antimicrobial clothing on clinical symptoms, quality of life, S. aureus colonization, AD medication use and the satisfaction regarding the clothing.

DETAILED DESCRIPTION:
This is a multi-center, double-blind, randomized controlled trial. Patients will be randomized in a 1:1:1 fashion to either therapeutic clothing without antimicrobial agents, antimicrobial therapeutic clothing based on chitosan or antimicrobial clothing based on silver for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Atopic dermatitis diagnosed according to the criteria of Williams (Williams 1994)
* Atopic dermatitis severity according to EASI at t = 0: > 6.0.

Exclusion Criteria:

* Treatment with oral antibiotics until 1 month before inclusion;
* Treatment with topical antibiotics until 1 week before inclusion;
* Treatment with systemic immunosuppressive agents or light therapy until 1 month before inclusion;
* Treatment with (antibacterial) therapeutic clothing until 1 month before inclusion;
* Impaired kidney function (anamnestic assessed)
* Pregnancy or pregnancy wish during study (anamnestic assessed)
* Hypersensitivity to silver (anamnestic assessed)
* Evidence of past non-compliance to treatments or appointment

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2020-03-17 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in the Eczema Area and Severity Index (EASI) | Two weeks for baseline, baseline, 1 month, 3 months 6 months and 12 months
  Change in disease severity measured by the EASI between the clothing without antimicrobial agents (control group) and microbial growth reducing/ antimicrobial clothing based on chitosan or silver (intervention groups) over 12 months. Minimum score is 0, maximum score is 72. A higher score indicates more sever eczema

SECONDARY OUTCOMES:
Change in global assessment of degree of impetiginisation | Baseline, 1 month, 3 months 6 months and 12 months
  Change in global assessment of degree of impetiginisation (pustules, oozing, crust formation) of dermatitis between the clothing without antimicrobial agents (control group) and microbial growth reducing/ antimicrobial clothing based on chitosan or silver (intervention groups), expressed as 0 - no impetiginisation, 1 - sporadic impetiginisation, 2 - mild impetiginisation, 3 - moderate impetiginisation, 4 - severe impetiginisation
Change in S. Aureus colonization | Baseline, 1 month, 3 months 6 months and 12 months
  Change in S. aureus colonization between the clothing without antimicrobial agents (control group) and microbial growth reducing/ antimicrobial clothing based on chitosan or silver (intervention groups) over 12 months
Change in the Patient Oriented Eczema Measure (POEM) | Baseline, 1 month, 3 months 6 months and 12 months
  Change in POEM or POEM for proxy completion in the case of children up to 10 years of age by their parents between the clothing without antimicrobial agents (control group) and microbial growth reducing/ antimicrobial clothing based on chitosan or silver (intervention groups) over 12 months. The POEM is a validated and standardized patient questionnaire.
Change in Patient global assessment (PGA) of disease severity | Baseline, 1 month, 3 months 6 months and 12 months
  Change in PGA severity of the disease between the clothing without antimicrobial agents (control group) and microbial growth reducing/ antimicrobial clothing based on chitosan or silver (intervention groups) over 12 months. This is a standardized patient questionnaire. The minimum score is 0, the maximum score is 4.
Change in the Dermatology Life Quality Index (DLQI) | Baseline, 1 month, 3 months 6 months and 12 months
  Change in DLQI between the clothing without antimicrobial agents (control group) and microbial growth reducing/ antimicrobial clothing based on chitosan or silver (intervention groups) over 12 months. Minimum score is 0, maximum score is 30. A higher score indicates more impact on quality of life. This outcome measure is assessed in patient >16 years old. The DLQI is a validated and standardized patient questionnaire.
Change in the Child Dermatology Life Quality Index (CDLQI) | Baseline, 1 month, 3 months 6 months and 12 months
  Change in CDLQI between the clothing without antimicrobial agents (control group) and microbial growth reducing/ antimicrobial clothing based on chitosan or silver (intervention groups) over 12 months. Minimum score is 0, maximum score is 30. A higher score indicates more impact on quality of life. This outcome measure is assessed in patient 4-16 years old. The CDLQI is a validated and standardized patient questionnaire.
Change in the Infant Dermatology Life Quality Index (IDLQI) | Baseline, 1 month, 3 months 6 months and 12 months
  Change in IDLQI between the clothing without antimicrobial agents (control group) and microbial growth reducing/ antimicrobial clothing based on chitosan or silver (intervention groups) over 12 months. Minimum score is 0, maximum score is 30. A higher score indicates more impact on quality of life. his outcome measure is assessed in patient <4 years old. The IDLQI is a validated and standardized patient questionnaire.
Change on the visual analogue scale (0-100 mm) for itch (VAS for itch) | Baseline, 1 month, 3 months 6 months and 12 months
  Change in degree of itching, expressed on a visual analogue scale (0-100 mm), between the clothing without antimicrobial agents (control group) and microbial growth reducing/ antimicrobial clothing based on chitosan or silver (intervention groups) over 12 months. Minimum score is 0, maximum score is 100mm. A higher score indicates more itch.
Change on the visual analogue scale (0-100 mm) for sleep disturbance (VAS for sleep disturbance) | Baseline, 1 month, 3 months 6 months and 12 months
  Change in degree of sleep disturbance, expressed on a VAS (0-100 mm), between the clothing without antimicrobial agents (control group) and microbial growth reducing/ antimicrobial clothing based on chitosan or silver (intervention groups) over 12 months. Minimum score is 0, maximum score is 100mm. A higher score indicates more sleep disturbance.
Change on the visual analogue scale (0-100 mm) for pain (VAS for pain) | Baseline, 1 month, 3 months 6 months and 12 months
  Difference in degree of pain, expressed on a VAS (0-100 mm), between the clothing without antimicrobial agents (control group) and microbial growth reducing/ antimicrobial clothing based on chitosan or silver (intervention groups) over 12 months. Minimum score is 0, maximum score is 100mm. A higher score indicates more pain.
Use emollients | Through study completion, 1 year
  Difference in emollients use between the clothing without antimicrobial agents (control group) and microbial growth reducing/ antimicrobial clothing based on chitosan or silver (intervention groups) is assessed weekly over 12 months. A patient questionnaire with two items (daily application frequency and number of days per week) will be used to assess this outcome.
Use of antibiotics | Through study completion, 1 year
  Difference in total use of antibiotics between the clothing without antimicrobial agents (control group) and microbial growth reducing/ antimicrobial clothing based on chitosan or silver (intervention groups) is assessed over 12 months. A weekly patient questionnaire with two items (dose and number of days) will be used to assess this outcome.
Use of topical corticosteroids | Through study completion, 1 year
  Difference in topical corticosteroid use between the clothing without antimicrobial agents (control group) and microbial growth reducing/ antimicrobial clothing based on chitosan or silver (intervention groups) is assessed over 12 months. A weekly patient questionnaire with two items (application frequency and number of days) will be used to assess this outcome.
Use of therapeutic clothing | Through study completion, 1 year
  Difference in therapeutic clothing use between the clothing without antimicrobial agents (control group) and microbial growth reducing/ antimicrobial clothing based on chitosan or silver (intervention groups) is assessed over 12 months. A weekly patient questionnaires with two items (number of nights worn and number of days worn) will be used to assess this outcome.
Quality-adjusted life year | Baseline, 1 month, 3 months 6 months and 12 months
  Difference in the QALYs based on EuroQol questionnaire between the clothing without antimicrobial agents (control group) and microbial growth reducing/ antimicrobial clothing based on chitosan or silver (intervention groups) over 12 months.
Recap of atopic eczema (RECAP) - a standardized questionnaire that measures (long term) AD control | Baseline, 1 month, 3 months, 6 months and 12 months
  Change in RECAP between the clothing without antimicrobial agents (control group) and microbial growth reducing/ antimicrobial clothing based on chitosan or silver (intervention groups) over 12 months. RECAP is an standardized instrument (patient questionnaire) with 10 items to measure (long-term) eczema control.
Dermatitis Family Impact (DFI) - a standardized questionnaire that measures the impact of a skin disease on the family of the patient | Baseline, 3 months, 6 months and 12 months
  Change in DFI on the family of the patient between the clothing without antimicrobial agents (control group) and microbial growth reducing/ antimicrobial clothing based on chitosan or silver (intervention groups) over 12 months. (only in patients <18 years). The minimum DFI score is 0 (= no impact on life of family). The maximum DFI score is 30 (= maximum effect on life of family). The DFI is a standerized patient questionnaire.
Family Dermatology Life Quality (FDLQI) - a standardized questionnaire that measures the impact of a skin disease on family members | Baseline, 3 months, 6 months and 12 months
  Change in FDLQI between the clothing without antimicrobial agents (control group) and microbial growth reducing/ antimicrobial clothing based on chitosan or silver (intervention groups) over 12 months. (by parents in patients <18 years, by partner in patients >18 years. This questionnaire assesses impairement of the quality of life of adult family members. A higher score indicates more impairment.
Parenting Stress Questionnaire | Baseline, 3 months, 6 months and 12 months
  Difference in parenting stress between the clothing without antimicrobial agents (control group) and microbial growth reducing/ antimicrobial clothing based on chitosan or silver (intervention groups) over 12 months. (Only in patients <18 years old). A T-score < 60 can be seen as normal, a higher score implicates clinical problems. The parenting stress questionnaire is a validated and standardized questionnaire
Quality of life (measured by the TAPCOL) | Baseline, 3 months, 6 months and 12 months
  Difference in quality of life between the clothing without antimicrobial agents (control group) and microbial growth reducing/ antimicrobial clothing based on chitosan or silver (intervention groups) over 12 months. The TAPCOL is validated and standardized questionnaire for children 6< years.
Quality of life (measured by the TACQOL ) | Baseline, 3 months, 6 months and 12 months
  Difference in quality of life between the clothing without antimicrobial agents (control group) and microbial growth reducing/ antimicrobial clothing based on chitosan or silver (intervention groups) over 12 months. The TAPQOL is a validated and standardized patient questionnaire for children (>5 years, <16 years)
Quality of life (measured by the TAAQOL ) | Baseline, 3 months, 6 months and 12 months
  Difference in quality of life between the clothing without antimicrobial agents (control group) and microbial growth reducing/ antimicrobial clothing based on chitosan or silver (intervention groups) over 12 months. The TAAQOL is a validated and standardized patient questionnaire for patients older than 16 years old.
Change of silver excretion in urine | Baseline, 1month, 3 months, 6 months and 12 months
  Difference in urinary silver excretion over time. Measured in the silver group only.

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne G.M.A Pasmans, Prof, Principal Investigator — Erasmus MC University Medical Center Rotterdam Dept Dermatology, Center of Paedatric Dermatology
Locations (1):
- Erasmus University Medical Center, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ragamin A, Fieten KB, Tupker RA, de Wit J, van Mierlo MMF, Jansen MS, Bronner MB, Schappin R, Schuren FHJ, Romeijn MLE, Arents BWM, Polinder S, de Graaf M, Rustemeyer T, Schuttelaar MLA, Pasmans SGMA. The effectiveness of antibacterial therapeutic clothing based on silver or chitosan as compared with non-antibacterial therapeutic clothing in patients with moderate to severe atopic dermatitis (ABC trial): study protocol for a pragmatic randomized controlled trial. Trials. 2021 Dec 11;22(1):902. doi: 10.1186/s13063-021-05836-y. PMID 34895292